CLINICAL TRIAL: NCT06738264
Title: Cardiovascular Risk Factors in Rheumatoid Arthritis Patients ( Comparison Between Seronegative and Seropositive Cases )
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amna Mohamed Mahmoud, resident doctor, Sohag University
Other Study IDs: Soh-Med--24-11-11MS
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- seronegative RA: Rheumatoid arthritis patients with negative rheumatoid factor and negative anti citrullinated proteins
- seropositive RA: Rheumatoid arthritis patients with positive rheumatoid factor and positive anti citrullinated proteins

SUMMARY:
The goal of this observational study is to learn about the long-term effects rheumatoid arthritis (RA) on cardiovascular system. The main question it aims to answer is:

Does seropositive raise risk of cardiovascular diseases more than seronegative RA ?

DETAILED DESCRIPTION:
We will investigate cardiovascular risk factors in patients with seronegative and seropositive rheumatoid arthritis.

Complete clinical examination including blood pressure (BP; using an automatic BP monitor) and heart rate (in beats per minute (bpm) either from an automatic BP monitor or a 12 lead ECG) will be measured according to the standard hospital procedures.

Routine Laboratory investigations, including complete blood count (CBC), Blood parameters, including autoantibodies and lipid profile will be determined), liver and kidney function tests, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), and lipid profile panel will be recorded.

The disease activity score-28 (DAS-28) and health assessment questionnaire (HAQ) will be assessed.

Framingham risk score will be calculated. Carotid doppler will be done . Current medications use including synthetic disease-modifying anti-rheumatic drugs (DMARDs), in addition to steroids, will be recorded.

Rheumatoid Factor and Anticitrullinated proteins antibodies presence will be determined.

Cardiovascular risk factors, including inflammation, hypertension, smoking, obesity, and dyslipidemia will be observed and a higher risk of Cardiovascular Diseases events (including myocardial infarction, stroke, and heart failure).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years.
* Both sexes.
* All patients with RA confirmed using the 2010 American College of Rheumatology/European Alliance of Associations for Rheumatology EULAR classification criteria
* RA diagnosed for at least six months to ensure chronicity.

Exclusion Criteria:

* Diagnosis of other significant autoimmune diseases (e.g., lupus, scleroderma).
* Use of medications known to significantly affect cardiovascular outcomes (e.g., certain anticoagulants or anti-inflammatory agents) that are not part of standard RA treatment.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: rheumatology outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
carotid artery wall thickness | one week
  abnormality in carotid doppler